CLINICAL TRIAL: NCT03453489
Title: Monitoring Telotristat Ethyl Inhibition of Tryptophan Hydroxylase (TPH) in Neuroendocrine Tumors Using ?-[11C]Methyl-L-tryptophan (AMT)-PET
Brief Title: AMT-PET in Monitoring Telotristat Etiprate Treatment in Participants With MetastaticNeuroendocrine Neoplasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-144; NCI-2018-00294 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-144 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH); 2017-144 (Other: Lexicon)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Carcinoid Syndrome; Metastatic Nonfunctional Well Differentiated Neuroendocrine Neoplasm
MeSH Terms: conditions — Serotonin Syndrome | interventions — alpha-methyltryptophan; Magnetic Resonance Spectroscopy; telotristat; telotristat ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (AMT-PET, telotristat etiprate) (Experimental): Participants undergo AMT-PET within 7 days prior to, and 9-14 days after start of telotristat etiprate treatment. Participants receive telotristat etiprate PO TID for 9-14 days.
  Interventions: Other: Carbon C 11 Alpha-methyltryptophan; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography; Drug: Telotristat Etiprate

INTERVENTIONS:
Other: Carbon C 11 Alpha-methyltryptophan — Undergo AMT-PET
  Other Names: 11C-alpha-methyltryptophan; 11C-AMT; [11C] AMT; alpha-[11C]methyl-L-tryptophan
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo AMT-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Drug: Telotristat Etiprate — Given PO
  Other Names: LX1032 Hippurate; LX1606; LX1606 Hippurate; TPH Inhibitor LX1606; Tryptophan Hydroxylase Inhibitor LX1032; Tryptophan Hydroxylase Inhibitor LX1606

SUMMARY:
This pilot trial studies how well telotristat etiprate works in treating participants with well differentiated neuroendocrine neoplasm that has spread to other places in the body and monitored by carbon C 11 alpha-methyltryptophan (AMT)-emission tomography (PET). Telotristat etiprate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Studying the changes within the tumor cells via AMT-PET may help doctors better understand how tumors respond to treatment with telotristat etiprate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of telotristat etiprate (telotristat ethyl) treatment in patients with advanced neuroendocrine tumors (NETs) using carbon C 11 alpha-methyltryptophan (alpha-[11C]methyl-?L-?tryptophan) (AMT)-?positron emission tomography (PET) as measured by changes in tumor maximum standardized uptake value (SUVmax).

SECONDARY OBJECTIVES:

I. Show that NETs will have increased AMT uptake on PET, as compared to surrounding non-tumor tissue at baseline.

II. Use compartmental modeling (in tumors with the left ventricle of the heart in the field-of-view) to measure change in AMT retention.

III. Measure change in AMT retention as mean standardized uptake value (SUVmean).

OUTLINE:

Participants undergo AMT-PET within 7 days prior to, and 9-14 days after start of telotristat etiprate treatment. Participants receive telotristat etiprate orally (PO) three times a day (TID) for 9-14 days.

After completion of study treatment, participants are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed, well-differentiated metastatic NETs
* Receiving stable-dose somatostatin analog (long-acting release [LAR], depot) for > 3 months before enrollment.
* Patients with 5-HIAA levels above or below the upper limit of normal range and those with unknown values at baseline are allowed to participate.
* Able to lie within the PET scanner for at least 70 minutes while undergoing scanning.
* ECOG performance status of 2 or better.
* Physical exam, CBC and Multiphasic (including electrolytes, BUN, creatinine, total bilirubin, AST, and ALT) must be done within 28 days of PET imaging and demonstrate adequate renal and liver function. Creatinine ≤ 2.5, total bilirubin ≤ 1.5 x upper limit of normal (ULN). AST and ALT ≤ 2.5 ULN.
* Patient must have a least one lesion greater than 2 cm on standard imaging (CT, MR, octreotide, or dotatate imaging within 8 weeks of the start of the study) that is judged amenable to AMT-PET.
* Women of child bearing potential must not be pregnant or breastfeeding. A negative urine or blood pregnancy test must be obtained in women with child bearing potential. Men and women with reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) on study entry and for the duration of study participation.
* Eligible and consent signed for imaging with AMT PET under protocol 2011-053.

Exclusion Criteria:

* Patients experiencing more than 12 watery bowel movements per day associated with volume contraction, dehydration, or hypotension, or showing evidence of enteric infection are excluded
* Patients are excluded if they had undergone tumor-directed therapy within 3 months
* Patients cannot be on a targeted agent (e.g., sunitinib or everolimus) or receiving cytotoxic chemotherapy (e.g., capecitabine or temozolomide); they cannnot be on telotristat ethyl; previous use is acceptable if the patient has been off for over one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Shields, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 61 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Achieved SUVmax Reduction of 20% or More Between Baseline and Follow up Scan
Description: The proportion of patients who achieved maximum standardized uptake value (SUVmax) reduction of 20% or more between baseline and follow up scan. It will be reported with a one-sided, 90% confidence limit.
Time Frame: Baseline up to follow up, assessed up to 3 months
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Number analyzed (Participants) | 4
Proportion of participants | 0 [0 to 1]

2. Secondary Outcome: Change in Mean Standardized Uptake Value (SUVmean)
Description: Will be reported as percent change with two-sided 95% confidence intervals. Paired t test will be used for pre-and post-treatment SUVs if normality assumption holds.
Time Frame: Baseline up to 3 months
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Number analyzed (Participants) | 4
Percentage change | 46.01 [-56.06 to 148.08]
Statistical Analysis 1: Comparison: Treatment (AMT-PET, Telotristat Etiprate); Test type: Other; p = 0.837, t-test, 2 sided

3. Secondary Outcome: Neuroendocrine Tumors Visibility
Description: Proportion of patients with visible neuroendocrine tumors at baseline out of total number of patients. The outcome will be reported as proportion and 95% CI
Time Frame: At baseline
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Number analyzed (Participants) | 4
Proportion of participants | 1 [0.51 to 1]

4. Secondary Outcome: Difference in SUVmax of AMT Uptake Between the Tumor Mass and Background at Baseline
Description: Difference will be reported as percent of (SUVmax.tumor - SUVmax.background)/SUVmax.background in the baseline scan with 95% Confidence Interval
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
Number analyzed (Participants) | 4
Percentage | 451.90 [271.21 to 632.60]

ADVERSE EVENTS:
Time Frame: From the date of informed consent until 4 weeks after the treatment completion, up to 3 months.
Arm/Group | Treatment (AMT-PET, Telotristat Etiprate)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03453489/Prot_SAP_000.pdf